CLINICAL TRIAL: NCT06433336
Title: Effect of Blood Pressure on Cardiovascular Outcomes and Recurrence After Catheter Ablation in Patients With Atrial Fibrillation
Acronym: AF BP
Status: Completed | Type: Observational
Sponsor: Lanzhou University Second Hospital (Other)
Responsible Party: Principal Investigator, Xiaowei Zhang, lanzhou university second hospital, Lanzhou University Second Hospital
Other Study IDs: lanzhou university second hosp; lanzhou university (Other: lanzhou university second hospital)
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation, Persistent; Blood Pressure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Effect of blood pressure on cardiovascular outcomes and recurrence after catheter ablation in patien: Atrial Fibrillation Recurrence Pulmonary Vein Isolation

SUMMARY:
Effect of blood pressure on cardiovascular outcomes and recurrence after catheter ablation in patients with atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were age >18 years and a diagnosis of AF by electrocardiogram during the preceding six months or on admission

Exclusion Criteria:

No follow-up

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Between February 2019 and December 2024, 800 consecutive patients who had been referred to lanzhou University second Hospital for treatment of AF and underwent successful ablation were assessed
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
cardiovascular events | 1 years
  death AMI stroke

CONTACTS AND LOCATIONS:
Overall Officials: xiao wei xiaowei zhang, PHD, Principal Investigator — Lanzhou University Second Hospital
Locations (1):
- Lanzhou University Second Hospital, Lanzhou, Gansu, China